CLINICAL TRIAL: NCT05527834
Title: VNRX-7145-104: an Open-label, Cross-over Study to Evaluate the Effect of Food on the Pharmacokinetics, Safety, and Tolerability of Ceftibuten/VNRX-7145 in Healthy Participants.
Brief Title: Food Effect on Ceftibuten/VNRX-7145 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VNRX-7145-104; 272201600029C-P00017-9999-1 (NIH)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ceftibuten

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 will assess the impact of a high fat meal.
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten
- Cohort 2 (Experimental): Cohort 2 will be conducted to assess the impact of an alternative lower fat meal if administration with high fat meal has a food effect on drug exposure.
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten
- Cohort 3 (Experimental): Cohort 3 will evaluate realistic fasting intervals and/or additional meal types if administration with food has a food effect on drug exposure.
  Interventions: Drug: VNRX-7145; Drug: Ceftibuten

INTERVENTIONS:
Drug: VNRX-7145 — Single oral dose
Drug: Ceftibuten — Single oral dose

SUMMARY:
This is an open label, two period (fasted and fed), crossover study in up to 3 cohorts of 12 healthy adult participants per cohort (up to 36 participants in total). The pharmacokinetics (PK) of the inactive prodrug VNRX-7145, its active parent drug VNRX-5236, and ceftibuten will be evaluated after a single oral dose of ceftibuten/VNRX-7145.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-65 years
* Males or non-pregnant, non-lactating females
* Body mass index (BMI): ≥18.5 kg/m2 and ≤32.0 kg/m2
* Laboratory values meeting defined entry criteria

Exclusion Criteria:

* History of drug allergy or hypersensitivity to penicillin, cephalosporin, or β-lactam antibacterial drug
* Conditions that potentially alter absorption and/or excretion of orally administered drugs
* Congenital or acquired immunodeficiency syndrome
* Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hr (predose) through 48 hours for fasting subjects and 0 hr (predose) through 72 hours for fed subjects
  Maximum observed plasma concentration (Cmax)
AUC0-t | 0 hr (predose) through 48 hours for fasting subjects and 0 hr (predose) through 72 hours for fed subjects
  Area under the plasma concentration-time curve (AUC) from time 0 up to the last quantifiable concentration at time t (AUC0-t)
AUC0-inf | 0 hr (predose) through 48 hours for fasting subjects and 0 hr (predose) through 72 hours for fed subjects
  AUC from time 0 extrapolated to infinity (AUC0-inf)

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Hamed, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- ICON Plc., Lenexa, Kansas, United States